CLINICAL TRIAL: NCT05391022
Title: A Phase 1, 2-Part Study to Evaluate the Effect of Food on Pharmacokinetics of Pelabresib (CPI-0610) and the Effect of Pelabresib on QTc in Patients With Advanced Malignancies
Brief Title: Study Evaluating Food Effect and QTc in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Constellation Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPI 0610-05; 2022-000896-38 (EudraCT Number); CDAK539A12106 (Other: Novartis)
Record Dates: First submitted 2022-05-05; First posted 2022-05-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignancies; Solid Tumor; Hematological Malignancy
Keywords: Pelabresib; CPI 0610
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Run-In Food Effect Period (Experimental): Unblinded, open label drug will be administered once in a fasted state and twice in a fed state with a minimum of 5 days between each dose prior to entering the continuous treatment phase.
  Interventions: Drug: Pelabresib
- Continuous Treatment Period (Experimental): Unblinded, open label drug will be administered once daily for 14 consecutive days followed by a 7 day break, which is considered 1 cycle of treatment (1 cycle = 21 days).
  Interventions: Drug: Pelabresib

INTERVENTIONS:
Drug: Pelabresib — Pelabresib monohydrate tablets
  Other Names: CPI 0610

SUMMARY:
Phase 1 2-part study to evaluate the effect of food on pharmacokinetics of pelabresib (CPI-0610) and the effect of pelabresib on QTc in patients with advanced malignancies

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Confirmed diagnosis of an advanced malignancy for which no effective standard treatment options are available
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2

Exclusion Criteria:

* Chronic or active conditions and/or concomitant medication use that would prohibit treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Run-In Food Effect Period: Area under the concentration time curve (AUC) based on pelabresib concentrations in plasma measured using validated plasma assay | 21 days
  The primary endpoint for the food effect is to investigate the effects high and low-fat meals have on the oral bioavailability of single doses of pelabresib
Run-In Food Effect Period: maximal plasma concentration (Cmax) based on pelabresib concentrations in plasma measured using validated plasma assay | 21 days
  The primary endpoint for the food effect is to investigate the effects high and low-fat meals have on the oral bioavailability of single doses of pelabresib
Run-In Food Effect Period: Time to maximal plasma concentration (Tmax) based on pelabresib concentrations in plasma measured using validated plasma assay | 21 days
  The primary endpoint for the food effect is to investigate the effects high and low-fat meals have on the oral bioavailability of single doses of pelabresib
Continuous Treatment Period: Changes in QT and QTc intervals | 12 months
  The primary endpoint of the QT portion is to determine the effect of single and multiple doses of pelabresib on QT/QTc prolongation

SECONDARY OUTCOMES:
-In Food Effect Period: Total amount (Ae[∞]) and fraction of dose (fe) of pelabresib | 24 hours
  Ae(∞) and fe of pelabresib excreted into urine
Run-In Food Effect Period and Continuous Treatment Period: incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs) | 12 months
  Safety: TEAEs and treatment-emergent SAEs

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - Gabrail Cancer Center Research, Canton, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Start Mountain Region, West Valley City, Utah
- Georgia (3):
  - Hight Technology Hospital Medcenter, Batumi
  - K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Simon Khechinashvili University Hospital, Tbilisi
- Spain (4):
  - Barcelona HM Nou Delfos, Barcelona
  - Madrid - FJD, Madrid
  - START CIOCC Hospital HM Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocío, Seville